CLINICAL TRIAL: NCT04164940
Title: A Multi-centre Registry Study on Patient Trajectories After Interventions for Alcohol-related Health Problems in Somatic Hospital Wards, for People in Late Adulthood (60+)
Brief Title: Patient Trajectories for Older Adults Admitted to Hospital for Alcohol-related Problems
Status: Recruiting | Type: Observational
Sponsor: Helse Stavanger HF (Other Government)
Collaborators: Helse Vest (Other); Helse Fonna (Other); Helse Møre og Romsdal HF (Other Government); Sorlandet Hospital HF (Other Government); Helse Sor-Ost (Other Government); Lovisenberg Diakonale Hospital (Other); Oslo University Hospital (Other); Vestre Viken Hospital Trust (Other)
Responsible Party: Sponsor
Other Study IDs: ID734
Record Dates: First submitted 2019-11-12; First posted 2019-11-15 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Alcohol Consumption; Alcohol; Harmful Use; Health Risk Behaviors; Alcohol Dependence
MeSH Terms: conditions — Alcohol Drinking; Health Risk Behaviors; Alcoholism | interventions — Ethanol; Methods

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Age 21-30: Patients aged 21-30 when admitted to hospital and receiving brief alcohol intervention
  Interventions: Other: Brief alcohol intervention
- Age 31-40: Patients aged 31-40 when admitted to hospital and receiving brief alcohol intervention
  Interventions: Other: Brief alcohol intervention
- Age 41-50: Patients aged 41-50 when admitted to hospital and receiving brief alcohol intervention
  Interventions: Other: Brief alcohol intervention
- Age 51-60: Patients aged 51-60 when admitted to hospital and receiving brief alcohol intervention
  Interventions: Other: Brief alcohol intervention
- Age 61-70: Patients aged 61-70 when admitted to hospital and receiving brief alcohol intervention
  Interventions: Other: Brief alcohol intervention
- Age 71-80: Patients aged 71-80 when admitted to hospital and receiving brief alcohol intervention
  Interventions: Other: Brief alcohol intervention
- Age 81 and older: Patients aged 81 and older when admitted to hospital and receiving brief alcohol intervention
  Interventions: Other: Brief alcohol intervention

INTERVENTIONS:
Other: Brief alcohol intervention — Brief alcohol intervention already implemented in daily routine by the individual hospitals.

SUMMARY:
Alcohol is contributing to many health problems and disorders, as well as accidents and social problems. Alcohol consumption has been on the rise the past 25 years, especially in Norway. The highest increase is found in older adults, in line with the development in most other countries in the western world. Older adults have a higher risk for alcohol related health problems, due to age related physiological changes, medical conditions and medications. Still, alcohol use is seldom addressed for older people. This means that older people rarely receive help to change alcohol habits.

Norwegian health authorities have issued mandates ordering the regional health trusts to implement strategies in somatic hospital wards, mental health services and drug treatment services to identify and treat alcohol and drug problems affecting the patients' health.

In this observational study we will explore patient trajectories three years prior to and three years after an admittance to hospital where risky or harmful alcohol consumption is identified and brief interventions are delivered. Hospitals that have implemented such strategies are invited to the study. Patient trajectories are studied in national health registries. This will provide important knowledge on what characterizes the patients identified, and what happens after they have received a brief intervention related to a hospital admittance.

DETAILED DESCRIPTION:
This is a multi-centre registry study in Norwegian medical and surgical hospitals. The project is focusing on patients aged 60+, receiving an intervention for alcohol-related health problems in somatic hospital wards in one year, and without a previous history of referral or treatment in specialized health care for an alcohol or drug problem. Other age groups of adults will be used as control groups. The included patients will also be their own control group, where we compare registry data on the trajectories three years following the alcohol intervention with registry data from the three years preceding the intervention.

The recruited hospitals will have different strategies for identification of and interventions for alcohol-related health problems, and the choice of methods is thus outside of our control. All inhabitants in Norway are registered with a personal identification number. This individual identifier makes the linkage between the participants and the different registries possible. Data from these registries will enable the study of serious incidents, as well as of diagnoses, medications and other treatments, welfare and benefits, and causes of death. Data will be gathered three years retrospectively and 3 years prospectively, related to the index hospital stay where alcohol is addressed and a brief intervention is delivered.

Inclusion criteria for patients are age 21+, no previous treatment history for drug or alcohol problems in specialized health care, admitted to medical or surgical hospital ward, identified risky or harmful alcohol consumption, accepting an alcohol intervention and accepting study participation. Baseline data collected are AUDIT C, question no 10 from the full AUDIT and classification of alcohol consumption (risky or harmful). All other variables are extracted from the national health registries (reimbursement data from primary health care and secondary health care, prescription database, Cause of death registry, Norwegian Trauma Registry and social security data, marital status, professional status).

ELIGIBILITY:
Inclusion Criteria:

* Age 21 or older, no previous alcohol use disorder or substance use disorder, admitted to hospital which has implemented screening and brief alcohol intervention strategies, written consent to participate

Exclusion Criteria:

* specialized treatment for alcohol use disorder og drug use disorder during the three years prior to recruitment

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 21 years or older admitted to medical or surgical hospital wards offering some kind of screening and brief alcohol intervention as part of the daily routine, and without a prior diagnosis of AUD or SUD.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-10-23 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Alcohol use disorder (AUD) | Three years
  Diagnosis of AUD after recruitment in the study
Prescriptions for AUD | Three years
  Prescriptions for the treatment of alcohol use disorder

SECONDARY OUTCOMES:
Health care | Three years
  Diagnoses and procedures in primary and secondary health care
Trauma | Three years
  Serious trauma registered in trauma registry
Death | Three years
  Death and cause of death
Prescriptions for addictive drugs | Three years
  Prescriptions for any drug with addictive potential

CONTACTS AND LOCATIONS:
Overall Officials: Torgeir G Lid, MD PhD, Principal Investigator — Helse Stavanger HF
Locations (1):
- StavangerUH, Stavanger, Norway

IPD SHARING:
Plan to Share IPD: No